CLINICAL TRIAL: NCT01191151
Title: Orthopaedic Sports Medicine, Arthroscopy, and Related Surgery Registry Using the Web-based OrthoIllustrated Surgical Outcomes System
Brief Title: Web Based Orthopaedic Sports Medicine Registry
Status: Terminated | Type: Observational
Why Stopped: Sponsor made buisness decision to close SOS Software, and terminate collecting data
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SOS #1
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Degenerative and Traumatic Pathology of the Knee; Degenerative and Traumatic Pathology of the Shoulder and Elbow; Degenerative and Traumatic Pathology of the Foot and Ankle; Degenerative and Traumatic Pathology of the Hand and Wrist; Degenerative and Traumatic Pathology of the Hip
Keywords: Orthopedic surgery; sports medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orthopedic injury, osteoarthritis: All eligible patients receiving orthopedic, sports medicine, arthroscopy and related surgery or nonoperative treatment

SUMMARY:
The purpose of this study is to establish an international, web based clinical registry to collect baseline characteristics of patients undergoing orthopaedic, sports medicine, arthroscopy, and related surgery, and the subsequent outcomes and cost-effectiveness associated with the surgical procedures and nonoperative treatments.

ELIGIBILITY:
Inclusion Criteria:

* All patients electing to schedule routine and medically indicated orthopedic, sports medicine, arthroscopy and related surgery or nonoperative treatment

Exclusion Criteria:

* Non English or Spanish speaking
* vulnerable populations, excluding minors

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort will be selected from clinic patients scheduling surgery or nonoperative treatment
Sampling Method: Non-Probability Sample
Enrollment: 12500 (Actual)
Dates: Start 2010-09; Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Change in pain | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Adams, MD, Principal Investigator — Arthrex, Inc.
Locations (258):
- United States (220):
  - Andrews Sports Medicine & Orthopedic Center, Birmingham, Alabama
  - Southern Orthopaedic Surgeons, Montgomery, Alabama
  - Alaska Hand-Elbow-Shoulder Surgical Specialists, Anchorage, Alaska
  - Steward Orthopedics and Sports Medicine, Phoenix, Arizona
  - The Orthopedic Clinic Association (Biocartilage), Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - The Orthopedic Clinic Association, Phoenix, Arizona
  - Arizona Bone and Joint Specialists, Scottsdale, Arizona
  - Agility Center, Bentonville, Arkansas
  - Adventist Health Bakersfield, Bakersfield, California
  - Los Angeles Institute of Foot and Ankle Surgery, Burbank, California
  - Blatz Orthopaedics and Sports Medicine, Campbell, California
  - PRISM, Campbell, California
  - Sierra Pacific Orthopedics, Fresno, California
  - Greater Long Beach Orthopaedics, Los Alamitos, California
  - USC Department of Orthopedic Surgery, Los Angeles, California
  - Kerlan Jobe Orthopaedic Clinic, Los Angeles, California
  - Mammoth Hospital, Mammoth Lakes, California
  - Premier Hip Arthroscopy, Marina del Rey, California
  - Orthomed Center, Modesto, California
  - Marin Orthopedic and Sports Medicine, Novato, California
  - Children's Hospital of Orange County, Orange, California
  - Congress Orthopaedic Associates, Pasadena, California
  - The Orthopedic Specialty Center of Northern California, Roseville, California
  - Sacramento Orthopedic Center, Sacramento, California
  - John G. Lane MD Inc., San Diego, California
  - Synergy Specialists Medical Group, San Diego, California
  - Advanced Orthopaedics and Sports Medicine Inc., San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - Anderson Knee and Shoulder Center, San Francisco, California
  - SBSPMA, San Francisco, California
  - Alta Orthopaedics, Santa Barbara, California
  - Orthopedic Surgical Practice, Santa Barbara, California
  - Children's Hospital Los Angeles, Santa Monica, California
  - Santa Monica Orthopedics and Sports Medicine Group, Santa Monica, California
  - Walnut Creek Orthopedics & Sports Medicine, Walnut Creek, California
  - Joint Preservation Institute, Walnut Creek, California
  - Muir Orthopaedic Specialists, Walnut Creek, California
  - Samimi Orthopedic Group, West Covina, California
  - Children's Hospital Colorado (BioCartilage), Aurora, Colorado
  - Boulder Institute for Sports Medicine, Boulder, Colorado
  - OrthoONE at Rose Medical Center, Denver, Colorado
  - Advanced Orthopedic and Sports Medicine Specialists, Denver, Colorado
  - Integrative Sports Medicine LLC, Fort Collins, Colorado
  - Panorama Orthopedic & Spine Center, Golden, Colorado
  - Steadman Hawkins Clinic, Greenwood Village, Colorado
  - BioLOGIC Regenerative Medicine, Steamboat Springs, Colorado
  - Orthopaedics of Steamboat Springs, Steamboat Springs, Colorado
  - Advanced Orthopedics New England, Bloomfield, Connecticut
  - ONS, Greenwich, Connecticut
  - First State Orthopaedics, Newark, Delaware
  - Morgan Kalman Clinic, Wilmington, Delaware
  - Washington Orthopaedics & Sports Medicine, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia
  - Medstar/Georgetown University, Washington D.C., District of Columbia
  - Ortho Stem Center, Aventura, Florida
  - Orthopaedic Surgery Associates, Boynton Beach, Florida
  - Coastal Orthopedics and Pain Management and Sports Medicine, Bradenton, Florida
  - North Tampa Orthopaedics & Sports Medicine, Brooksville, Florida
  - National Training Center, Sports Medicine Institute, Clermont, Florida
  - UHZ Sports Medicine Institute, Coral Gables, Florida
  - Joint Implant Surgeons of Florida, Fort Myers, Florida
  - Andrews Orthopaedic & Sports Medicine Center, Gulf Breeze, Florida
  - Advanced Shoulder Orthopaedics, Jupiter, Florida
  - First Choice Medical Group, Melbourne, Florida
  - OrthoMiami, Miami, Florida
  - Collier Sports Medicine, Naples, Florida
  - Frank McCormick MD, Pompano Beach, Florida
  - Orthopaedic Associates of St. Augustine, Saint Augustine, Florida
  - Florida Orthopedic Foot & Ankle Center, Sarasota, Florida
  - Tallahassee Orthopedic Clinic (Mejia), Tallahassee, Florida
  - Champions Orthopedics, Augusta, Georgia
  - Harbin Clinic, Rome, Georgia
  - Atlanta Orthopaedic Institute, Stockbridge, Georgia
  - Valdosta Orthopedic Associates, Valdosta, Georgia
  - Humphrey Shoulder Clinic, Eagle, Idaho
  - Suburban Orthopaedics, Bartlett, Illinois
  - Midwest Orthopedics at Rush, Chicago, Illinois
  - Center for Athletic Medicine, Chicago, Illinois
  - Fox Valley Orthopaedic Institute, Geneva, Illinois
  - MK Orthopaedics, Surgery and Rehabilitation, Joliet, Illinois
  - Illinois Bone and Joint Institute, Libertyville, Illinois
  - Advanced Orthopedic and Spine Care, Oak Lawn, Illinois
  - Midwest Orthopaedic Consultants, Orland Park, Illinois
  - Skyline Orthopedics, Orland Park, Illinois
  - American Health Network, Avon, Indiana
  - Southern Indiana Orthopedics, Columbus, Indiana
  - Central Indiana Orthopedics, Muncie, Indiana
  - Henry Community Orthopaedics and Sports Medicine, New Castle, Indiana
  - KUMC, Kansas City, Kansas
  - Orthopaedic and Sports Medicine Consultants, Leawood, Kansas
  - Mid-America Orthopedics, Wichita, Kansas
  - Advanced Orthopaedic Associates, Wichita, Kansas
  - King's Daughters Medical Center, Ashland, Kentucky
  - Medical Center Bowling Green Clinic, Bowling Green, Kentucky
  - BlueGrass Orthopedics, Lexington, Kentucky
  - Ochsner Sports Medicine Institute, Jefferson, Louisiana
  - Louisiana State University, Kenner, Louisiana
  - Lafayette General Orthopaedic Center, Lafayette, Louisiana
  - Louisiana Orthopaedic Specialists, Lafayette, Louisiana
  - Coastal Orthopedics & Sports Medicine, Brunswick, Maine
  - OA center for Orthopedics, Portland, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - Maryland Sports Medicine Center, Olney, Maryland
  - Potomac Valley Orthopaedic Associates, Chartered, Olney, Maryland
  - Peninsula Orthopaedic Assoc., Salisbury, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Ortho.Boston, Needham Heights, Massachusetts
  - Orthopedic Care Physician Network, North Easton, Massachusetts
  - Boston Sports & Shoulder Center, Waltham, Massachusetts
  - Ortho Michigan, Flint, Michigan
  - River Valley Orthopedics, Grand Rapids, Michigan
  - West Michigan Orthopedics, Grand Rapids, Michigan
  - Mid-Michigan Orthopaedic Institution, Lansing, Michigan
  - Motor City Orthopedics and Sports Medicine Institute, Novi, Michigan
  - Ascension Medical Group, Rochester Hills, Michigan
  - Michigan Center for Regenerative Medicine, Rochester Hills, Michigan
  - Heartland Orthopedic Specialists, Alexandria, Minnesota
  - Summit Orthopedics, Maplewood, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Columbus Orthopaedic Clinic, Columbus, Mississippi
  - Mississippi Sports Medicine, Jackson, Mississippi
  - Rush Foundation Hospital, Meridian, Mississippi
  - Starkville Orthopedic Clinic, Starkville, Mississippi
  - Orthopedic Surgeons Inc, Blue Springs, Missouri
  - Regeneration Orthopedics, Chesterfield, Missouri
  - The Orthopedic Center of St. Louis, Chesterfield, Missouri
  - St. Peters Bone & Joint, City of Saint Peters, Missouri
  - Columbia Orthopedic Group, Columbia, Missouri
  - Missouri Orthopaedic Institute, Columbia, Missouri
  - Advanced Orthopedic & Sports Medicine dba Sano, Lee's Summit, Missouri
  - Bluetail Medical Group, St Louis, Missouri
  - Motion Orthropaedics, St Louis, Missouri
  - Bridger Orthopaedic and Sports Medicine, Bozeman, Montana
  - Desert Orthopaedic Center, Las Vegas, Nevada
  - Total Sports Medicine, Las Vegas, Nevada
  - Lourdes Medical Assoc., Burlington, New Jersey
  - North Jersey Orthopaedic Clinic, Glen Rock, New Jersey
  - Mercer-Bucks Orthopaedics, Lawrence, New Jersey
  - Seaview Orthopedics, Ocean City, New Jersey
  - Skyview Orthopedic Associates, Sparta, New Jersey
  - New Mexico Orthopaedic Associates, Albuquerque, New Mexico
  - Las Cruces Orthopaedic Associates, Las Cruces, New Mexico
  - Taos Orthopaedic Institute, Taos, New Mexico
  - Capital Region Orthopaedics, Albany, New York
  - Excelsior Orthopaedics, LLP, Amherst, New York
  - SUNY Downstate Health Sciences University, Brooklyn, New York
  - Mount Sinai Medical Center, New York, New York
  - NY Orthopedics, New York, New York
  - Oneida Health, Oneida, New York
  - Manhattan Orthopedic Care, Staten Island, New York
  - Regional Orthopedics, Staten Island, New York
  - Asheville Orthopedic Associates, Asheville, North Carolina
  - Southeastern Sports Medicine & Orthopedics, Asheville, North Carolina
  - EmergeOrtho, Asheville, North Carolina
  - Appalachian Regional, Boone, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - OrthoCarolina, Charlotte, North Carolina
  - The Cleveland Shoulder Institute #2, Beachwood, Ohio
  - Adena Bone & Joint Center, Chillicothe, Ohio
  - Beacon Orthopaedics and Sports Medicine LTD, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - The Cleveland Shoulder Institute, Cleveland, Ohio
  - OhioHealth Orthopedic Surgeons, Columbus, Ohio
  - Toledo Orthopaedic Surgeons, Toledo, Ohio
  - Orthopedic Foot and Ankle Center, Worthington, Ohio
  - Oklahoma Sports Science and Orthopedics, Oklahoma City, Oklahoma
  - Southern Oregon Orthopedics, Medford, Oregon
  - Oregon Orthopedic & Sports Medicine Clinic, LLP, Oregon City, Oregon
  - Sports Medicine Oregon, Tigard, Oregon
  - Coordinated Health, Allentown, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - Temple Orthopaedics and Sports Medicine, Philadelphia, Pennsylvania
  - Burke and Bradley Orthopedics, Pittsburgh, Pennsylvania
  - UPMC-St. Margarets Hospital, Pittsburgh, Pennsylvania
  - So County Orthopaedics, Wakefield, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - McLeod Health, Florence, South Carolina
  - CNOS, Dakota Dunes, South Dakota
  - Bone and Joint Institute of Tennessee, Franklin, Tennessee
  - Tennessee Orthopaedic Clinics, Knoxville, Tennessee
  - OrthoKnox, Knoxville, Tennessee
  - Aubrey Smith Orthopedics, Amarillo, Texas
  - Austin Sports Medicine, Austin, Texas
  - Texas Institute for Hip & Knee Surgery, Austin, Texas
  - Austin Shoulder Institute, Austin, Texas
  - Texas Orthopedic Specialists, PLLC, Bedford, Texas
  - Texas Health, Fort Worth, Texas
  - Craig Ranch Orthopaedics, Frisco, Texas
  - Fondren Orthopedic Group, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Laredo Sports Medicine Clinic, Laredo, Texas
  - Center for Orthopedic Surgery, Lubbock, Texas
  - TTUHSC Department of Orthopedics, Lubbock, Texas
  - West Texas Orthopedics, Midland, Texas
  - Children's Health, Plano, Texas
  - OSSMSA, San Antonio, Texas
  - The San Antonio Orthopaedics Group, San Antonio, Texas
  - The San Antonio Orthopaedic Group, San Antonio, Texas
  - Sterling Ridge Orthopaedics & Sports Medicine, Spring, Texas
  - Azalea Orthopedics, Tyler, Texas
  - Advent Healthcare, Waco, Texas
  - Waco Orthopedic & Sports Medicine Clinic, Waco, Texas
  - Heiden Orthopedics, Salt Lake City, Utah
  - Center of Orthopedic & Rehabilitation Excellence, West Jordan, Utah
  - Mansfield Orthopaedics, Waterbury, Vermont
  - Anderson Clinic, Arlington, Virginia
  - G2 Orthopedics and Sports Medicine, Glen Allen, Virginia
  - National Sports Medicine Institute, Lansdowne Town Center, Virginia
  - Advanced Orthopedics, Richmond, Virginia
  - Atlantic Orthopaedic Specialists, Virginia Beach, Virginia
  - Virginia Institute for Sports Medicine, Virginia Beach, Virginia
  - Orthopedics International, Kirkland, Washington
  - The Sports Medicine Clinic, Seattle, Washington
  - Weirton Medical Center, Weirton, West Virginia
  - Prevea Health, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
- Canada (4):
  - Fortius Sport & Health, Burnaby, British Columbia
  - Durham Sports Specialists, Ajax, Ontario
  - Pinnacle Health Sciences, Richmond Hill, Ontario
  - Jason Smith Medical Corporation, Scarborough Village, Ontario
- Caribbean Shoulder and Elbow Institute, San Juan, Puerto Rico
- South Africa (19):
  - Alberlito Hospital, Ballitoville
  - NMK Orthopaedics, Berea
  - Sports Science Institute of South Africa, Cape Town
  - Gateway Private Hospital, Durban
  - Hillcrest Private Hospital, Durban
  - Inkosi Albert Luthuli Hospital, Durban
  - Life Entabeni Hospital, Durban
  - Mediclinic Howick, Howick
  - Walk A Mile Centre For Advanced Orthopaedics, Lyttelton
  - Greenacres Hospital, Newton Park
  - Maritzburg Orthopaedic Centre, Northdale
  - Maritzburg Orthopaedic Centre, Pietermaritzburg
  - Drs Beekarun Moodley Rajah And Partners, Pinetown
  - Cape Shoulder Institute, Plattekloof
  - Netcare Moot Hospital, Rietfontein
  - Centre for Sports Medicine and Orthopaedics, Rosebank
  - Center for Sports Medicine & Orthopaedics, Rosebank
  - Umhlanga Medical Centre, Umhlanga
  - Westville Hospital, Westville
- United Kingdom (14):
  - Martyn Snow, Birmingham, West Midlands
  - BMI Clementine Churchill Hospital, Middlesex
  - Surrey Orthopaedic Clinic, Ottershaw
  - NDORMS, Oxford
  - Poole Hospital, Poole
  - Circle Hospital, Reading
  - Southampton University Hospital, Southampton
  - Mackay Orthopaedic Associates, Stirling
  - MacKay Orthopaedic Associates, Stirling
  - University Hospital of North Tees, Stockton-on-Tees
  - Walsall Manor Hospital, Walsall
  - Wrightington Hospital, Wigan
  - The Windsor Knee Clinic, Windsor
  - Windsor Knee Clinic, Windsor

REFERENCES:
- [Background] Gliklich RE, Dreyer NA, editors. Registries for Evaluating Patient Outcomes: A User's Guide. 2nd edition. Rockville (MD): Agency for Healthcare Research and Quality (US); 2010 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK49444/ PMID 21204321
- [Background] Schemitsch EH, Bhandari M, Boden SD, Bourne RB, Bozic KJ, Jacobs JJ, Zdero R. The evidence-based approach in bringing new orthopaedic devices to market. J Bone Joint Surg Am. 2010 Apr;92(4):1030-7. doi: 10.2106/JBJS.H.01532. No abstract available. PMID 20360530
- [Background] Capozzi JD, Rhodes R. Examining the ethical implications of an orthopaedic joint registry. J Bone Joint Surg Am. 2010 May;92(5):1330-3. doi: 10.2106/JBJS.I.01410. PMID 20439699